CLINICAL TRIAL: NCT03670199
Title: Improving the Quality of Life of Cancer Patients Through a Perioperative and Coordinated Nutrition and Physical Care Program.
Acronym: PENDICOQ
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 6117
Record Dates: First submitted 2018-07-11; First posted 2018-09-13 (Actual); Last update posted 2021-09-13 (Actual); Status verified 2021-09

CONDITIONS: Undernourished; Digestive Cancer
MeSH Terms: conditions — Malnutrition; Gastrointestinal Neoplasms | interventions — Nutrition Assessment; Diet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): nutritional and functional management coordinated by dieticians and physiotherapists, with adapted nutritional and physical advice and support, realized with the use of Nutrimus booklet in order to facilitate coordination and delivration of cares proposed to the patients
  Interventions: Other: Dietary intervention; Other: Intensify physiotherapist intervention
- Control group (Active Comparator): usual preoperative advice for patients who undergoing surgical procedure concerning nutritional cares and physical activity
  Interventions: Other: Dietary advice; Other: Physiotherapist intervention

INTERVENTIONS:
Other: Dietary advice — Nutritional status assessment Explanation of standard nutritional advices with an written explanation sheet
  Arms: Control group
Other: Physiotherapist intervention — Respiratory capacity Functional capacity
  Arms: Control group
Other: Dietary intervention — Nutritional status assessment Presentation of the Nutrimus booklet by the coordinating dietitian Establishment or adaptation of a nutritional support (prescription of nutritional supplements if necessary). Delivery and explanation of the preoperative nutritional counseling support
  Arms: Experimental group
Other: Intensify physiotherapist intervention — Respiratory capacity Functional capacity Tips adapted for physical activity and strengthening or maintenance of muscle mass Presentation of respiratory physiotherapy exercises to prevent postoperative bronchial congestion Nutrition and physical mobilization tips with the Nutrimus booklet
  Arms: Experimental group

SUMMARY:
Hospitalization, for cancer patients, exposes to a risk of undernutrition which has the effect of significantly increasing infections, pressure ulcers, muscle wasting, loss of autonomy, impaired function and delayed healing.

All of these factors contribute to increase the length of stay in hospital, thus lengthening the spiral of undernutrition, which has serious consequences for the patient welbeing, health establishments and public health.

Undernutrition has been the subject of many studies over the last twenty years, that outline that an adequate nutritional management exerts a direct effect on the reduction of comorbidities and duration of hospitalization.

However, there are periods, in the preoperative course of care, where nutritional and phisical care are not realized in the current clinical practice whereas they could be done, for example, between the diagnosis and the consultation of anesthesia, between the anesthesia consultation and the surgical procedure and the end of hospitalization of the patient.

Current management is usually limited to the period of hospitalization which tends to be reduced. This situation is reinforced by the absence of relays at home, dietary consultations being not reimbursed by French health insurance.

Moreover, a preliminary survey, conducted in 2012 during the pre-operative outpatient anesthesia consultation, shows that 26% of patients are already clinically malnourished, with 16.5 % of them who have lost more than 10% of their weight.

DETAILED DESCRIPTION:
Then, the investigators hypothesize that the combination of perioperative nutrition and mobilization program coordinated andrealized by dieticians and physiotherapists, with the Nutrimus follow-up booklet, would improve the post-operative evolution of patients and reduce their postoperative comorbidities.

This management, initiated at the consultation of anesthesia, would include an accurate nutritional diagnosis, nutritional and physical support therapy to improve their nutritional and muscular status.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 18 years old
* Patient with Karnofsky index superior or equal to 60%.
* Patient with cancer of the following digestive tract: peritoneal carcinoma, sarcoma, pancreas, rectum, esophagus, stomach diagnosed or under diagnosis
* Patient admitted for a scheduled surgery at least 10 days after a preoperative consultation
* Patient affiliated to a social health insurance scheme
* Patient having dated and signed an informed consent
* Patient having been informed of the results of the prior medical examination

Exclusion Criteria:

* Inhospital patients
* Patient admitted in emergency
* Impossibility of giving the patient information (alteration of patient's cognitive function)
* Illiteracy or dyscalculia
* Patients protected (guardianship, curatorship, safeguard of justice)
* Pregnancy, breastfeeding
* Subject in exclusion period (determined by a previous or ongoing study),
* Patient included in another ongoing clinical trial
* Patient with neuro-endocrine cancer
* Patient reoperated for the same pathology

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-01-29 (Actual); Primary Completion 2024-04-28 (Estimated); Study Completion 2024-04-28 (Estimated)

PRIMARY OUTCOMES:
Variation of the Medical Outcome Study Short Form 36 score | Change in score at 30 days before surgery and 1 Day before hospital discharge
  Use of a scale for quality of life

SECONDARY OUTCOMES:
Sarcopenia index measurement | 30 days before surgery
  Measure from routine preoperative Computerized Tomography scan
Satisfaction score of the Nutrimus tool | 6 months postoperative
  Use of a questionnaire
Ease of use of the Nutrimus tool | 6 months postoperative
  Use of a questionnaire
Measurement of the Medical Outcome Study Short Form 36 score | Change in score at 1 day before surgery, 1 day before the end of hospitalization, 1 Month, 3 Months and 6 Months post hospitalization
  Use of a scale for quality of life
Evaluation of nutritional parameters | Change in values measures at 30 days to 10 days, 1 day before surgery, 1 day before the end of hospitalization, 1 Month, 3 Months and 6 Months post hospitalization
  Use of a notebook
Evaluation of respiratory and functional capacities | Change in measures at 30 days to 10 days, 1 day before surgery, 1 day before the end of hospitalization, 1 Month, 3 Months and 6 Months post hospitalization
Pain assessment | Change in score at 30 days to 10 days, 1 day before surgery, 1 day before the end of hospitalization, 1 Month, 3 Months and 6 Months post hospitalization
  Use of a visual analogue scale Measure of score from 0 to 10
Length hospitalization | Duration (in days) of patient's hospitalization
  Length (in days) between hospital admission and discharge

CONTACTS AND LOCATIONS:
Overall Officials: Alain PARDIGNAC, Principal Investigator — Strasbourg Universitary hospitals
Locations (1):
- Service de Médecine Interne et Nutrition, Hôpital de Hautepierre, Hôpitaux universitaires de Strasbourg, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No